CLINICAL TRIAL: NCT03864887
Title: Optical Assessment on Brain Death Via a Multiple-phase Protocol at Varied Fraction of Inspired O2
Brief Title: Optical Assessment on Brain Death Via a Oxygen Supply Procedure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ting Li, Professer, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: Brain Death of AMS
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Brain Death
Keywords: Brain death; Oxygen metabolism; Near infrared spectroscopy
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Brain death patients for HLH Oxygen: Brain-dead patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of high-low-high procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of high-low-high procedure; Device: Optical monitor for hemodynamic parameter.
- Brain death patients for LHL Oxygen: Brain-dead patients were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of low-high-low procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of low-high-low procedure; Device: Optical monitor for hemodynamic parameter.
- Healthy people for HLH Oxygen: Healthy people were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of high-low-high procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of high-low-high procedure; Device: Optical monitor for hemodynamic parameter.
- Healthy people for LHL Oxygen: Healthy people were supplied with oxygen at varied FIO2 at medical premised range.The protocol is Oxygen supply of low-high-low procedure. During the procedures, the Δ[Hb] and Δ[HbO2] time courses were collected by Optical monitor for hemodynamic parameter.
  Interventions: Procedure: Oxygen supply of low-high-low procedure; Device: Optical monitor for hemodynamic parameter.

INTERVENTIONS:
Procedure: Oxygen supply of high-low-high procedure — The protocol consisted of 1-hour resting, 3-minute baseline measurement, half-hour measurement at 60% FIO2 (phase I, high oxygen), half-hour measurement at 40% FIO2 (phase II, low oxygen) and half-hour measurement at 60% FIO2 (phase III, high oxygen).
  Groups: Brain death patients for HLH Oxygen; Healthy people for HLH Oxygen
Procedure: Oxygen supply of low-high-low procedure — The protocol consisted of 1-hour resting, 3-minute baseline measurement, half-hour measurement at 40% FIO2 (phase I, low oxygen), half-hour measurement at 60% FIO2 (phase II, high oxygen) and half-hour measurement at 40% FIO2 (phase III, low oxygen).
  Groups: Brain death patients for LHL Oxygen; Healthy people for LHL Oxygen
Device: Optical monitor for hemodynamic parameter. — Near infrared spectroscopy probes of tow wavelengths were attached on the subjects' foreheat to detect the changes of hemodynamic parameters.

SUMMARY:
This study aims to evaluate brain death with optical probes. The changes of hemodynamic parameters including oxyhemoglobin (HbO2) and deoxyhemoglobin (Hb) were detected by near infrared spectroscopy probes attached on the forehead of patients. A multiple-phase protocol at varied fraction of inspired O2 were utilized during the assessment.

DETAILED DESCRIPTION:
Brain death is an irreversible loss of all brain functions, and the assessment is crucial for organ supply for transplantation. The noninvasive, sensitive, universally available and timely ancillary method to assess brain death has not been established. This study aims to evaluate brain death with optical probes. The changes of hemodynamic parameters including oxyhemoglobin (HbO2) and deoxyhemoglobin (Hb) were detected by near infrared spectroscopy probes attached on the forehead of patients. A multiple-phase protocol at varied fraction of inspired O2 were utilized during the assessment. The concentration changes ratios of oxyhemoglobin to deoxyhemoglobin (Δ[HbO2]/Δ[Hb]) in the cerebral cortex of brain-dead patients were significantly higher than those of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had brain death or serious brain trauma.
* Healthy people who are interested in optical assessment of hemodynamic parameters

Exclusion Criteria:

* Patients who are in pregnancy or have plan to conception.
* Patients who have vertebra surgery or have plan of surgery.
* Patients who are inappropriate to join this trial judged by the radiologists or specialists.

  * AIDS, Active Hepatitis, Tuberculosis, Syphilis
  * Patients who regularly take anticoagulants, antiplatelet drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals of any gender. Mostly hired in the City of Tianjin, P.R.China
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Δ[HbO2] | 1 day during the whole experiment
  The changes of oxyhemoglobin concentrations in prefrontal cortex.
Δ[Hb] | 1 day during the whole experiment
  The changes of deoxyhemoglobin concentrations in prefrontal cortex.

SECONDARY OUTCOMES:
Heart rate | 1 day during the whole experiment
  Heart rate of patient recorded by bed-side physiological monitor.
Blood pressure | 1 day during the whole experiment
  Blood pressure of patient recorded by bed-side physiological monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- NIRS assessment for brain death, Tianjin, Tianjin Municipality, China